CLINICAL TRIAL: NCT02344667
Title: Randomized Feasibility Study of Stereotactic Body Radiotherapy (SBRT) for Localized Prostate Cancer: Cyberknife vs. Volume Modulated Arc Therapy
Brief Title: Feasibility Study of Stereotactic Body Radiotherapy (SBRT) for Localized Prostate Cancer: Cyberknife vs. VMAT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Juravinski Cancer Center (Other)
Collaborators: Juravinski Cancer Centre Foundation (Other)
Responsible Party: Principal Investigator, Dr. Himu Lukka, Professor, Juravinski Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RD-157
Record Dates: First submitted 2015-01-13; First posted 2015-01-26 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2015-01

CONDITIONS: Prostatic Neoplasms
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cyberknife (Experimental): Cyberknife based SBRT 36.25 Gy in 5 fractions
  Interventions: Radiation: Stereotactic Body Radiotherapy
- Volume Modulated Arc Therapy (Experimental): Volume Modulated Arc Therapy based SBRT 36.25 Gy in 5 fractions
  Interventions: Radiation: Stereotactic Body Radiotherapy

INTERVENTIONS:
Radiation: Stereotactic Body Radiotherapy

SUMMARY:
Recent studies support the use of Stereotactic Body Radiation Therapy (SBRT) for the treatment of localized prostate cancer (PrCa). SBRT is a way to deliver radiation very precisely allowing higher doses to be delivered with fewer treatments, potentially improving patient outcomes. Cyberknife and Volume Modulated Arc Therapy (VMAT) are accepted SBRT techniques. However, the effects of the specific SBRT treatment technique on patient outcomes have not been evaluated in randomized trials.

Although such a trial would be of great interest, patients' willingness to participate is unclear. Multiple patient and clinician factors contribute to the decision to enter a randomized trial. This feasibility study will evaluate patients' willingness to participate in a trial comparing Cyberknife and VMAT SBRT for the treatment of early stage PrCa. Patients accepting enrolment will be randomized to one of the two types of SBRT delivery. Up to 66 patients will be approached, and up to 40 randomized. A questionnaire will help to identify the factors influencing the patient's decision to participate or not. This study will gather information on feasibility, PSA control, patient outcomes and side effects, and will inform the design of a future randomized phase II/III study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of adenocarcinoma of the prostate
* Histological evaluation of prostate biopsy with assignment of a Gleason score to the biopsy material; Gleason scores ≤ 7
* Clinical stage T1-2b (AJCC 7th edition)
* PSA ≤ 10 ng/mL. PSA should not be obtained within 10 days after prostate biopsy.
* ECOG Performance Status 0-1

Exclusion Criteria:

* Prior or concurrent invasive malignancy (except non-melanomatous skin cancer) or lymphomatous/hematogenous malignancy unless continually disease free for a minimum of 5 years.
* Evidence of distant metastases
* Regional lymph node involvement
* Previous radical surgery (prostatectomy), cryosurgery, or HIFU for prostate cancer. Previous pelvic irradiation, prostate brachytherapy, or bilateral orchiectomy
* Previous hormonal therapy, such as LHRH agonists or LHRH antagonists, anti-androgens, estrogens, or surgical castration
* Use of finasteride or dutasteride within 30 days prior to registration. PSA should not be obtained prior to 30 days after stopping finasteride or dutasteride.
* Previous or concurrent cytotoxic chemotherapy for prostate cancer
* Age < 18
* Patient unable to provide study-specific informed consent
* Inability to complete the Expanded Prostate Cancer Index Composite (EPIC) questionnaire

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-03; Primary Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Patient acceptability of a randomized trial comparing Cyberknife and Volume Modulated Arc Therapy (VMAT) based SBRT techniques for the treatment of localized prostate cancer as measured by number of patients willing to participate in randomized trial. | 15 months